CLINICAL TRIAL: NCT01053377
Title: A Randomised Controlled Trial on the Effect of Post-exposure Oseltamivir Prophylaxis on Influenza Transmission in Nursing Homes
Acronym: PEPpIE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Institute for Public Health and the Environment (RIVM) (Other Government)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Marianne van der Sande, Institute of Public Health and the Environment
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL27938.041.09
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2009-12

CONDITIONS: Influenza
Keywords: Influenza; Tamiflu; Osteltamivir; Transmission; Prevention; Resistance; Post-Exposure Profylaxe
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamiflu (Active Comparator)
  Interventions: Drug: Tamiflu (verum)
- Placebo Tamiflu (Placebo Comparator)
  Interventions: Drug: Tamiflu placebo

INTERVENTIONS:
Drug: Tamiflu (verum)
  Arms: Tamiflu
Drug: Tamiflu placebo
  Arms: Placebo Tamiflu

SUMMARY:
The incidence of severe morbidity and mortality following an influenza infection during the annual influenza epidemics is highest among the elderly population and 90% of influenzaassociated mortality occurs in this group. Vaccination is considered the best preventive intervention available but offers only partial protection. The protective effect decreases with advancing age and existing co-morbidity. Therefore, in spite of high compliance with vaccination, the risk of influenza-related complications among nursing-home residents, is particularly high, and consequently also the associated disease and economic burden. There is debate on the potential health benefit of the antiviral activity of oseltamivir as an effective supplementary intervention to prevent or contain influenza outbreaks in nursing homes. Although effectiveness of post-exposure prophylaxis (PEP) with oseltamivir on preventing transmission has been demonstrated in trials among healthy (mainly unvaccinated) adults and children, effectiveness has not yet been assessed among vulnerable vaccinated highrisk groups, such as the elderly population in nursing homes. If proven (cost)effective, oseltamivir could have considerable benefits in this setting, although constraints relating to implementation need to be addressed as well.

DETAILED DESCRIPTION:
Objective If proven (cost)effective, without inducing antiviral resistance, oseltamivir could have considerable benefits in this setting, although constraints relating to implementation need to be addressed as well. If not (cost)effective if this fragile population, resources can be better spent on other activities to support nursing home residents.

Study design:

A randomised controlled trial on the effect of PEP with oseltamivir versus placebo on transmission of influenza in nursing homes, linked to virological monitoring of possible development of resistance and impact on transmission and outcome, linked with a cost effectiveness analysis, and an exploration of logistical and ethical issues which could interfere with successful implementation.

Study population:

This trial will be nested in the recently established Network of Nursing Homes (SNIV). SNIV has been initiated and is coordinated by the RIVM Centre of Infectious Disease Control. Baseline data on the population in these nursing homes is already routinely collected, and epidemiological and virological surveillance of ILI/influenza is established, in collaboration with the local laboratories.

Intervention:

Post-exposition prophylaxis with oseltamivir or placebo. Once laboratory confirmation has been obtained in an index case, all residents of that implicated unit only will be randomly assigned to PEP with either oseltamivir 75 mg or placebo once daily for 10 days. Data on co-morbidity, medication and other potential confounders for susceptibility to a clinical influenza infection will be collected prior to the start of PEP. The index patient (and any secondary patients) will be treated therapeutically with oseltamivir. Main study parameters/endpoints: Transmission, the primary trial outcome measurement, is defined as a newly laboratory confirmed influenza in the same unit 12 hours or more after the start of PEP. Assuming 30 homes participate, that annually 30% of nursinghomes experience a confirmed influenza outbreak in on average two units, than we can recruit 20 units per season. Assuming that without effective prophylaxis ongoing transmission occurs in 40% of the units, we will have at least 80% power after 3 seasons with a two-sided alpha=0.05 to demonstrate a reduction in transmission of 70%.

Furthermore, this trial offers an excellent opportunity to evaluate the possible emergence of resistance against oseltamivir if used under such circumstances, by analysing the occurrence of viral mutations under oseltamivir therapy (for index- and for any secondary cases). In addition, we will assess the relative cost-effectiveness of PEP with oseltamivir per nursing home unit, compared to not using PEP by prospectively collecting information on the number of influenza infections and related complications, duration of symptoms, use of medical services by secondary cases, as well as sickness leave of staff.

Finally, potential ethical and logistical restrictions for the large scale use of oseltamivir will be documented prospectively.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Burden and risks of this trial will be minimal, as we will not deviate from current standing practices, in which some nursing homes offer PEP and others don't, following the diagnosis of influenza on a unit.

ELIGIBILITY:
Exclusion Criteria:

* Kidney dialyses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Transmission of influenza from person to person | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Public Health and the Environment, Bilthoven, Utrecht, Netherlands

REFERENCES:
- See also: Research site — http://www.peppieonderzoek.nl